CLINICAL TRIAL: NCT04078386
Title: A Phase II Study of RC18, a Recombinant Human B Lymphocyte Stimulator Receptor:Immunoglobulin G( IgG ) Fc Fusion Protein for Injection for the Treatment of Subjects With Primary Sjögren's Syndrome
Brief Title: A Study of TACI-antibody Fusion Protein Injection (RC18) in Subjects With Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18C012
Record Dates: First submitted 2019-07-18; First posted 2019-09-06 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Primary Sjögren's Syndrome
MeSH Terms: interventions — RC-18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RC18 240mg (Experimental)
  Interventions: Biological: RC18 240 mg
- RC18 160 mg (Experimental)
  Interventions: Biological: RC18 160 mg
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Patients received the test group Placebo weekly administered subcutaneously for 24 times.
  Arms: Placebo
Biological: RC18 240 mg — Arm Description:Patients received the test group RC18 240mg weekly administered subcutaneously for 24 times.
  Arms: RC18 240mg
Biological: RC18 160 mg — Patients received the test group RC18 160mg weekly administered subcutaneously for 24 times.
  Arms: RC18 160 mg

SUMMARY:
The purpose of this study is to initially observe the safety and effectivity of RC18 in Participants with Primary Sjögren's Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent ;
* Patient with primary Sjögren's syndrome according to the European - American consensus group criteria.
* Seropositive at screening for anti-Ro/Sjögren's syndrome type A(SSA) antibodies
* ESSDAI score ≥ 5.

Exclusion Criteria:

* Diagnosis of secondary Sjogren's syndrome, such as rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis and other autoimmune diseases;
* Abnormal laboratory parameters need to be excluded, including but not limited to:
* Immunosuppressive agents were used within 4 weeks prior to randomization.;
* The use of hydroxychloroquine was allowed during the trial, and the pre-randomized drug regimen was stable for less than 12 weeks;
* Use of biological agents for targeted therapy in the first 6 months of randomization;
* Treatment of primary Sjogren's syndrome with traditional Chinese medicine and proprietary Chinese medicine within 4 weeks before randomization;
* The use of saliva-stimulating drugs within 7 days prior to randomization;
* Sodium hyaluronate eye drops, artificial tears can be used, and the stability time of the randomized pre-medication scheme is less than 4 weeks;
* Intravenous immunoglobulin therapy or plasma exchange therapy within 6 months before randomization;
* Infection with herpes zoster or HIV and hepatitis C virus(HCV) antibody positive;
* Currently suffering from active hepatitis or severe liver lesions and history;
* Malignant tumor patients ;
* Combined with involvement of important organs or neuropathy;
* Have participated in any clinical trial in the first 28 days of the initial screening or 5 times half-life period of the study compound (taking the time for the shorter).
* Pregnant , lactating women and men or women who have birth plans during the research;
* Investigator considers candidates not appropriating for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
The amount of change of European League Against Rheumatism Sjögren's syndrome disease activity(ESSDAI) score compared to the baseline at week 24. | week 24
  ESSDAI= European League Against Rheumatism Sjögren's syndrome disease activity index score.The ESSDAI includes It includes 12 domains (ie, organ systems: cutaneous,respiratory, renal, articular, muscular，peripheral nervous system (PNS), central nervous system (CNS), haematological, glandular,constitutional,lymphadenopathic,biological).. Each domain is divided into 3-4 levels of activity.The higher the score, the more serious the symptoms ,that is,the worse the results.Subscales are combined by summed.

SECONDARY OUTCOMES:
The amount of change of ESSDAI score compared to the baseline at week 12. | week 12
  ESSDAI= European League Against Rheumatism Sjögren's syndrome disease activity index score.The ESSDAI includes It includes 12 domains (ie, organ systems: cutaneous,respiratory, renal, articular, muscular，peripheral nervous system (PNS), central nervous system (CNS), haematological, glandular,constitutional,lymphadenopathic,biological).. Each domain is divided into 3-4 levels of activity.The higher the score, the more serious the symptoms ,that is,the worse the results.Subscales are combined by summed.
The amount of change of European League Against Rheumatism Sjögren'sSyndrome Patient Reported Index(ESSPRI) score compared to the baseline at week 12 and week 24 | week 12，24
  European League Against Rheumatism Sjögren's Syndrome Patient Reported Index.Dryness, pain, somatic and mental fatigue were identified as the main symptoms of patients with primary SS. It was suspected that a single 0-10 numerical scale for each domain was sufficient to assess these symptoms.The higher values represent a worse outcome.Subscales are combined by averaged.
Doctors assess overall changes in disease activity relative to baseline at week 12 and week 24 | week 12,24
  The measurement tool is Visual Analogue Scale/Score（VAS）.The doctor assesses participant's disease activity on a VAS of 0 - 100 mm on the questionnaire form.
Overall patient assessment of disease activity compared to baseline at week 12 and week 24 | week 12,24
  The measurement tool is Visual Analogue Scale/Score（VAS）. The participant assesses his/her own disease activity on a VAS of 0 - 100 mm on the questionnaire form.
Changes in short form(SF)-36 relative to baseline at week 12 and week 24 | week 12,24
  SF-36=36-item short form. As a concise health questionnaire, SF-36 summarized the quality of life of the subjects from eight aspects: physiological function, physical pain, general health condition, energy, social function, emotional function and mental health.The SF-361 is a self-report, 36 item survey measuring health-related quality-of-life. Thirty-five items are used to construct 8 scales. An additional item measures health transition.The higher values represent a better outcome.Subscales are combined by averaged.
Statistical Analysis of the variation of multidimensional fatigue inventory relative to baseline at week 12 and week 24 | week 12,24
  Multidimensional Fatigue Inventory.The MFI is a 20-item scale designed to evaluate fi ve dimensions of fatigue: general fatigue, physical fatigue, reduced motivation,reduced activity, and mental fatigue.The higher values represent a worse outcome,Subscales are combined by summed.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Remegen,Ltd., Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu D, Fang J, Zhang S, Huang C, Huang C, Qin L, Li X, Chen M, Liu X, Liu Y, Li Z, Hu J, Bao C, Wei W, Tian J, Duan X, Zeng X. Efficacy and safety of telitacicept in primary Sjogren's syndrome: a randomized, double-blind, placebo-controlled, phase 2 trial. Rheumatology (Oxford). 2024 Mar 1;63(3):698-705. doi: 10.1093/rheumatology/kead265. PMID 37399108